CLINICAL TRIAL: NCT04806139
Title: Translation of an Evidence-based Exercise Program for Remote Delivery to Rural, Older Cancer Survivors
Brief Title: Survivors Taking Action With Remote Exercise Training
Acronym: JumpSTART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Nancy Gell, Associate Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UVMCC 2100/CHRMS 00001375
Record Dates: First submitted 2021-03-08; First posted 2021-03-19 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Cancer
Keywords: physical activity; rural; cancer; older adults
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: The intervention will be offered to two groups (goal sample size of 15 participants in each group, with additional recruiting to account for attrition). The second Remote Enhance Fitness group will begin following the completion of the first group.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group - Remote Enhance Fitness (Experimental): Participants assigned to the intervention group will participated in a 16-week remote exercise intervention. Following a home/space environment and technology needs assessment, participants will attend a one-on-one orientation and practice class with a research assistant. Participants will join a live-streamed, instructor-led group Enhance Fitness exercise session for 1-hour, 3 days/week for 4 months (16-weeks).
  Interventions: Behavioral: Remote Enhance Fitness
- Waitlist Control (No Intervention): Participants randomized to the waitlist control group will be offered the opportunity to participate in the Remote Enhance Fitness class after study measures are completed. Cuff weights will be provided along with technical orientation, support, and equipment as needed.

INTERVENTIONS:
Behavioral: Remote Enhance Fitness — The Remote Enhance Fitness Intervention will include live-streamed exercise classes (1-hour long, 3 days per week, 16 weeks). Certified Enhanced Fitness trainers will lead the exercise classes per Enhance Fitness guidelines, including modifications and gradual progression. During weeks 8-12 participants will have the option to wear a Fitbit during classes for up to 6 class session (2 weeks) for collection of heart rate, steps, and physical activity intensity along with ratings of perceived exertion (RPE) during exercise classes.
  Arms: Intervention Group - Remote Enhance Fitness

SUMMARY:
The proposed pilot study will test the acceptability and feasibility of a sixteen-week, two-arm randomized control physical activity intervention in older cancer survivors. The Survivors Taking Action with Remote exercise Training (JumpSTART) program is intended for cancer survivors (Stage I-III) age 60 or older, living in rural areas. The goal of this intervention is to increase physical activity opportunities for cancer survivors who are geographically isolated by offering exercise classes (EnhanceFitness) online. The real-time instruction of group-based classes helps older adults to exercise by establishing relationships, fostering social support and receiving corrective and supportive feedback from instructors that enhance self-efficacy for exercise.

ELIGIBILITY:
Inclusion Criteria:

* Rural residence by self-report and confirmed with Rural-Urban Commuting Area Codes
* Stage I-III cancer history
* Completion of adjuvant chemotherapy, radiation therapy, or surgery for cancer diagnosis
* Age 60 years or older
* Ability to walk for exercise
* Self-reported minimal or inconsistent participation in strengthening exercise and physical activity (< 150 minutes/week moderate-to-vigorous physical activity; confirmed with baseline accelerometer measures)
* Clearance for exercise based on a modified, combined Screening Cancer Survivors for Unsupervised Moderate-to-Vigorous Intensity Exercise and the Screening for Physical Activity Readiness Questionnaire (PAR-Q) or physician approval as needed based on the pre-screening/PAR-Q responses

Exclusion Criteria:

* Not available for the study duration
* Unable to communicate by phone
* Unable to attend exercise class at schedule time (M,W,F, time TBD)
* Currently enrolled in another exercise program
* Unable to communicate in English

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Patient Reported Outcome Measurement System (PROMIS)-Physical Function10a | 4 months
  Physical function will be assessed with the PROMIS Physical Function short form. This measure has 10 items and been validated for use in multiple populations including cancer survivors and people with multiple chronic conditions. Scale range is 1-5 (not at all, very much) with higher scores indicating worse physical function.
Fatigue | 4 months
  The Patient Reported Outcome Measurement System (PROMIS)-29 will be collected which includes 4 items on fatigue. Scale range is 1-5 (Not at all, Very much). Higher scores indicate worse fatigue
Sleep disturbance | 4 months
  The Patient Reported Outcome Measurement System (PROMIS)-29 will be collected which includes 4 items on sleep disturbance. Scale range is 1-5 (Never, Always). Higher scores indicate worse sleep disturbance.
Physical Activity (PA) and Sedentary Time Assessment | 4 months
  Physical activity and sedentary time will be assessed using the activPAL accelerometer. Participants will wear the device for seven (7) days during each measurement period. Overall PA levels will be assessed via daily step counts and minutes of moderate-to-vigorous physical activity and will be summed across the week. Accelerometer data will also include sedentary time and light physical activity time.

SECONDARY OUTCOMES:
Five time sit-to-stand test | 4 months
  Measure of strength (power): Score is in seconds with higher scores indicating worse physical performance. This assessment will be conducted remotely over video-conference.
30 second-sit-to-stand test | 4 months
  Strength (endurance) will be assessed using the validated 30 second sit-to-stand test: Score is in seconds with higher score indicating better physical performance. This assessment will be conducted remotely over video-conference.
Four-stage balance test | 4 months
  Measure of balance: Score is in seconds with completion of all 4 stages indicated better balance. This assessment will be conducted remotely over video-conference.
Duke Activity Status Index | 4 months
  Status will be assessed using a 12-item questionnaire that assesses the ability to do self-care, housework, sports, and other activities. Response options are "Yes" or "No" for each of the 12 items. Higher scores indicate higher functional fitness levels.
Technology Use and Acceptance | 4 months
  The 14-item short version of the Senior Technology Acceptance Model (STAM) has demonstrated reliability and validity to measure technology-related attitudinal beliefs, control beliefs, and anxiety in older adults. Scale is 1-10 with higher scores indicating higher technology use and acceptance.
Adapted Technology Acceptance Model Scale | 4 months
  The 10-item adapted version of the Technology Acceptance Model (TAM) has demonstrated reliability and validity to measure technology-related ease of use, usefulness, financial cost, and intention to use. Scale range is 1-7 (Strongly disagree to Strongly agree) and higher scores indicate better usability, usefulness, and more intention to use.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Gell, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No